CLINICAL TRIAL: NCT03990493
Title: A Study to Evaluate the Safety and Efficacy of PV-001-DV in Combination With Infusion of PV-001-DC in Patients With Advanced Melanoma
Brief Title: Intratumoral Injection of PV-001-DV Plus DC in Patients With Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PrimeVax Immuno-Oncology Inc. (Industry)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PV001-001 (Arm 3)
Record Dates: First submitted 2019-06-12; First posted 2019-06-19 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Advanced Melanoma

STUDY DESIGN:
Intervention Model Description: Single Group Assignment with Dose Modification
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PV-001-DV in Combination with PV-001-DC (Experimental): Intratumoral injection of PV-001-DV (1 injection) and IV Infusion of PV-001-DC (every 3 weeks for total of 4 infusions)
  Interventions: Biological: Dengue Virus-1 #45AZ5 (PV-001-DV); Biological: Autologous Monocyte-derived Lysate Pulsed Dendritic Cells (PV-001-DC)

INTERVENTIONS:
Biological: Dengue Virus-1 #45AZ5 (PV-001-DV) — Intratumoral injection of PV-001-DV (1 injection)
Biological: Autologous Monocyte-derived Lysate Pulsed Dendritic Cells (PV-001-DC) — IV Infusion of PV-001-DC (every 3 weeks for total of 4 infusions)

SUMMARY:
The purpose of this arm of the study is to evaluate the safety of PV-001-DC (autologous monocyte-derived dendritic cells pulsed with tumor lysate) when given in combination with PV-001-DV (Dengue Virus-1 strain #45AZ5) at the dose levels that were identified in the prior 2 arms and to determine if the combination can treat advanced melanoma.

Patients will have a prescribed amount of PV-001-DV injected into one of their melanoma tumors. Patients will go to the clinic and have a needle placed in a vein. The PV-001-DC product will be infused into the patient's vein. Approximately every 3 weeks, for a total of 4 treatments, patients will receive additional infusions of PV-001-DC Patients will be at the clinic for at least 1 hour following the end of each PV-001-DC infusion and if they feel fine, they may go home.

Approximately 49 days after the first infusion, patients will have a scan to see if their tumors have changed in size. Other scans may be performed during the study at different times. Patients will also have their blood and small samples of tumors tested for changes to the immune system. After 365 days, the trial will be completed for that patient.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy confirmed patients with un-resectable American Joint Committee on Cancer (AJCC), Stage III or IV melanoma who have measurable disease. Measurable disease is required, and is defined as tumor can be measured in one dimension along the longest diameter
2. Patients must have tumors that are not responsive having completed prior therapy with a Progressive Death (PD)-1 / PD-Ligand-1 (PDL-1), antagonist alone or in combination with anti-Cytotoxic T Lymphocyte Antigen 4 (CTLA-4). If the patient is positive for BRAF, the patient must have progressed on at least one BRAF inhibitor in addition to a PD-1 / PD-L1 inhibitor alone or in combination with CTLA4 for metastatic melanoma
3. Patients must be progressing after having completed one standard of care therapy for metastatic melanoma
4. Tumor specimens must be available for tumor lysates and immunological studies.
5. Tumors must be available for intratumoral injection of dengue virus. This includes cutaneous and subcutaneous lesions with ultrasound-guided injection.
6. Eastern Cooperative Oncology Group (ECOG), Performance Status of ≤ 2 (corresponds to a Karnofsky Performance Status (KPS) of ≥ 70).
7. Patients must be 18 years or older and able to give informed consent.
8. Adequate bone marrow function of White Blood Cell (WBC) count to ≥ 1,500/microliter (uL); platelet count ≥ 100,000/mm3; absolute neutrophil count (ANC) > 1,500/mm3
9. Patients must have adequate renal function by serum creatinine of ≤ 2.0 milligrams/decaliter (mg/dL).
10. Adequate hepatic function of bilirubin ≤ 2.5 mg/dL; Serum Glutamic Oxaloacetic acid Transaminase/ Serum Glutamic Pyruvic Transaminase (SGOT/SGPT) < 3× upper limit of normal (ULN).
11. Patients must have the required wash out periods from prior therapy:
12. Topical therapy: 2 weeks.
13. Chemotherapy and radiotherapy: 4 weeks.
14. Other investigational therapy: 4 weeks
15. Patients of reproductive potential and their partners must agree to use an effective (>95% reliability) form of contraception during the study and for 4 weeks following the last study drug. Patients who become pregnant during the course of the study will be withdrawn from the trial.
16. Women of reproductive potential must have a negative urine pregnancy test.
17. Patients should have a life expectancy of > 4 months.
18. Patient should be able to comply with the treatment schedule and have the ability to understand and the willingness to sign the informed consent document.
19. Patients with manageable Central Nervous System (CNS), metastases may be selected to this trial. CNS metastasis patients are eligible if the CNS metastases have had no progression for at least 4 weeks (as defined by Magnetic Resonance Imaging [MRI]/Computerized Tomography [CT]).

Exclusion Criteria:

1. Patients with positive antibody to any Dengue Virus serotype by tetravalent ELISA assay.
2. Patients with prior vaccinations or positive Ab detected by ELISA to: West Nile, St. Louis Encephalitis, or Yellow Fever
3. Pre-existing autoimmune or antibody mediated disease including systemic lupus erythematous, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, but excluding controlled thyroid disease, or the presence of autoantibodies without clinical autoimmune disease.
4. Known history of human immunodeficiency virus (HIV) or any active immunosuppressive systemic infection or a suppressed immune system, including acquired immuno-deficiency syndrome (AIDS) or HIV positivity and known hepatitis B or C infections (HCV or HBC), as assessed by serology.
5. Patients on immunosuppressive therapy. Concurrent steroid use of not more than an equivalent of 10 mg of prednisone is allowed.
6. Any other open wounds.
7. Previous organ transplantation.
8. Patients with clinically significant dermatological disorders, as judged by the clinical investigator (e.g., eczema or psoriasis), any skin lesions or ulcers, any history of atopic dermatitis, or any history of Darier's disease (Keratosis Follicularis).
9. Patients with White Blood Cell count <1,500/uL; platelet count <100,000/mm3; absolute neutrophil count (ANC) 1,500/mm3 (Grade 2)
10. Patients with inadequate renal function by serum creatinine of >1.5 x ULN (Grade 2)
11. Patients with inadequate liver function by SGPT/SGOT > 3x ULN, and bilirubin >2.5 mg/dl (Grade 2)
12. Patients with active infection or with a fever >101°F (38.5°C) within 3 days prior to the first scheduled treatment.
13. Concurrent participation in other treatment related clinical studies. Non-treatment studies (e.g. observation or tumor cell analysis studies) are allowed.
14. Prior malignancy (active within 3 years of screening) except basal cell or completely excised non-invasive squamous cell carcinoma of the skin, or in situ squamous cell carcinoma of the cervix.
15. Significant cardiovascular disease (i.e., New York Heart Association (NYHA) class 3 congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias).
16. Female patients who are pregnant or lactating.
17. Patients taken off Checkpoint Blockade agents: Ipilimumab, Nivolumab, Pembrolizumab, for Grade 3 or greater autoimmune toxicity. [7]
18. Patients who are positive for B-RafV600 mutation and are responding to targeted therapy.
19. Any other medical history, including laboratory results, deemed by the investigator to be likely to interfere with his/her participation in the study, or to interfere with the interpretation of the results.
20. Patients with endocrinopathy greater than grade III.
21. Patients who have undergone a splenectomy in their previous medical history will be excluded from this trial. Evidence of a splenectomy will be from history or records.
22. Prior history or serologic evidence of other flavivirus infections (yellow fever, St. Louis encephalitis, West Nile virus)
23. Prior history of having received a flavivirus vaccine
24. Patients who are actively taking Non Steroid Anti Inflammatory Drugs (NSAID) including aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events | 365 days
  Treatment-Emergent Adverse Event Incidence of patients receiving intratumoral injection of PV-001-DV in combination with IV infusion of PV-001-DC

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 365 days
  Tumor response will be measured per investigator's assessment according to RECIST v1.1 and iRECIST
Progression-Free Survival (PFS) | 365 days
  The length of time during the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse, up to the end of the study
Overall Survival (OS) | 365 days
  Overall Survival is measured from the date of enrollment to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date, up to the end of the study

IPD SHARING:
Plan to Share IPD: Undecided